CLINICAL TRIAL: NCT00778206
Title: PKUDOS: Phenylketonuria (PKU) Demographic, Outcomes, and Safety Registry
Acronym: PKUDOS
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: PKUDOS-01; PKUDOS Registry (Registry Identifier: PKUDOS)
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Phenylketonuria; Hyperphenylalaninaemia
Keywords: Phenylketonuria; Hyperphenylalaninemia; PKU; Phenylalanine
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. PKUDOS Registry: Patients with a confirmed diagnosis of Phenylketonuria (PKU) with hyperphenylalaninemia who have either received Kuvan therapy, or currently receive Kuvan therapy, or intend to begin receiving Kuvan therapy within 90 days of entering the registry.
- 2. PKU MOMS Subregistry: Patients with PKU who are pregnant at enrollment in the registry or who become pregnant while participating in the registry.
  Interventions: Drug: Kuvan

INTERVENTIONS:
Drug: Kuvan — -Recommended post-partum Assessments include: collection of baby's plasma at Birth, 1 Month and 6 months, and collection of mother's plasma and expressed breast milk sample at 1 Month.
  Other Names: sapropterin dihydrochloride
  Groups: 2. PKU MOMS Subregistry

SUMMARY:
The objective of this study is to evaluate the safety of long-term treatment with Kuvan.

DETAILED DESCRIPTION:
The PKUDOS program is a voluntary, multicenter, strictly observational program for patients with PKU who have either received Kuvan therapy, or currently receive Kuvan, or intend to begin receiving Kuvan therapy within 90 days of entering the registry.

ELIGIBILITY:
PKUDOS Registry

Inclusion Criteria:

* Patient has confirmed diagnosis of PKU with hyperphenylalaninemia documented by a Phenylalanine level of greater than or equal to 360 umol/L (6 mg/dL)
* Patient has previously received Kuvan
* Patient is currently receiving Kuvan
* Patient intends to receive Kuvan therapy within 90 days of enrollment into the registry
* The Patient is being followed at a PKUDOS participating center
* Willing and able to provide written authorization or, if under the age of 18 years, provide written assent (if required) and written patient authorization by a parent or legal guardian
* Willing to provide personal health information

Exclusion Criteria:

* Patients are not eligible to participate in PKUDOS if they are participating in a BioMarin-sponsored clinical study of Kuvan
* Patients not previously treated with Kuvan and patients that are unwilling to begin Kuvan therapy within 90 days of entry into the registry

PKU MOMS Subregistry

Inclusion Criteria:

* Willing to enroll in (or are already enrolled in) PKUDOS
* Agree to follow the standard of care for pregnant women with PKU in the United States (NIH, 200, NIH Consensus Statement)
* Agree to be followed by a hospital or PKU clinic offering the standard of care for maternal PKU
* Are within 10 weeks of their last menstrual period

Exclusion Criteria:

* Patients who have not adhered to the standard of care for pregnant women with PKU in the United States are not eligible to participate in PKU MOMS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of Phenylketonuria with hyperphenylalaninemia
Sampling Method: Non-Probability Sample
Enrollment: 1887 (Actual)
Dates: Start 2008-09; Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Observational Data Only | 15 years
  Registry data including demographic and baseline characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Lindstrom, MD, Study Director — BioMarin Pharmaceutical
Locations (45):
- United States (45):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - LAC and USC Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Diego, San Diego, California
  - Stanford University, Pediatrics, Stanford, California
  - Children's Hospital, University of Colorado School of Medicine, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami, Miller School of Medicine, Department of Human Genetics, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Tampa Children's Hospital, St. Joseph's Pediatric Endocrine Associates, Tampa, Florida
  - Emory University, Decatur, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wesley Pediatric Faculty Clinic, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Tulane University Medical School, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Children's Hosptial of Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - AHS Hospital Corp, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - University of Rochester Medical Center, Rochester, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State, Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christophers Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - West Virginia Genetics Center, Department of Pediatrics, Morgantown, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin